CLINICAL TRIAL: NCT06951204
Title: Evaluation of the Role of Genicular Nerve Block When Combined With Adductor Canal Block for Pain Control Following Knee Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FMASU MS170/2024
Record Dates: First submitted 2025-03-06; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-03

CONDITIONS: Post Operative Pain Control
Keywords: Genicular nerve block; Adductor canal block; motor sparing analgesia
MeSH Terms: interventions — Single Person

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adductor canal block (ACB) only (Active Comparator): This group will receive Adductor canal block only (control group)
  Interventions: Procedure: Adductor Canal Block (ACB) Only
- Adductor canal block (ACB) combined with Genicular nerve block (GNB) (Active Comparator): This group will receive Adductor canal block and Genicular nerve block
  Interventions: Procedure: Adductor canal block (ACB) combined with Genicular nerve block (GNB)

INTERVENTIONS:
Procedure: Adductor Canal Block (ACB) Only — All patients will receive adductor canal block under complete aseptic conditions using a high-frequency ultrasound guidance (Sonosite turbo M, Bothell, Washington,USA ). while patient is laying supine lower limbs will slightly abducted at the hips and flexed at the knees , using linear ultrasound probe(2.5-7.5MHZ) on the anterior aspect of the patient's thigh, At the level of mid-thigh, by moving probe medially until the boat shaped Sartorius muscle is visualized , at which the adductor canal is identified beneath the sartorius muscle, 20ml bupivacaine (0.25%) will be injected in the canal after a careful negative aspiration. The spread of the drug lateral and around the femoral artery will be seen real time on ultrasound
  Arms: Adductor canal block (ACB) only
Procedure: Adductor canal block (ACB) combined with Genicular nerve block (GNB) — All patients will receive adductor canal block as described above under complete aseptic conditions then they will receive the genicular nerve block using a high-frequency ultrasound guidance (Sonosite turbo M, Bothell, Washington,USA ), genicular nerve block will be done at three locations, i.e., superomedial, superolateral, and inferomedial locations of the condyle-shaft junction, while patient is lying supine linear ultrasound probe(2.5-7.5MHZ) will be used to target the superomedial, superolateral, and inferomedial genicular nerves,2ml bupivacaine (0.25%) will be injected in the 3 mentioned points after a careful negative aspiration
  Arms: Adductor canal block (ACB) combined with Genicular nerve block (GNB)

SUMMARY:
The intervention tests the efficacy of Genicular nerve block when combined with Adductor canal block in comparison with Adductor canal block alone to control post operative pain in knee arthroscopy

DETAILED DESCRIPTION:
A. Preoperative settings:

All patients will be assessed preoperatively by careful history taking, full physical examination, and laboratory evaluation. An informed written consent will be taken from every patient just before the surgery.

Intraoperative and postoperative settings:

On arrival to the operating room, baseline parameters such as ECG, mean arterial blood pressure, heart rate, and oxygen saturation will be recorded. Intravenous line will be inserted, and IV Ringer's solution will be started, then induction of general anesthesia: Preoxygenation with 100% oxygen will be carried out for 2-3 minutes. Induction of anesthesia will be done using intravenous fentanyl 1-2 µg/kg and propofol 1-2 mg/kg. Endotracheal intubation will be facilitated with atracurium 0.4-0.5 mg/kg. Proper intubation will be confirmed by ETCO2 and bilateral auscultation of the chest. Anesthesia will be maintained with 60:40 oxygen mixed with air and isoflurane 1.2%. Lungs will be ventilated using volume-controlled ventilation with tidal volumes and respiratory rate adjusted to maintain end tidal CO2 at 35-40 MMGH.

After induction of general anesthesia and intubation:

Group A: • All patients will receive adductor canal block under complete aseptic conditions using a high-frequency ultrasound guidance (Sonosite turbo M, Bothell, Washington, USA ). while patient is laying supine lower limbs will slightly abducted at the hips and flexed at the knees , using linear ultrasound probe(2.5-7.5MHZ) on the anterior aspect of the patient's thigh, At the level of mid-thigh, by moving probe medially until the boat shaped Sartorius muscle is visualized , at which the adductor canal is identified beneath the sartorius muscle, a, 20ml bupivacaine (0.25%) will be injected in the canal after a careful negative aspiration. The spread of the drug lateral and around the femoral artery will be seen real time on ultrasound.

Group B: All patients will receive adductor canal block as described above under complete aseptic conditions then they will receive the genicular nerve block using a high-frequency ultrasound guidance (Sonosite turbo M, Bothell, Washington, USA ), genicular nerve block will be done at three locations, i.e., superomedial, superolateral, and inferomedial locations of the condyle-shaft junction, while patient is lying supine linear ultrasound probe(2.5-7.5MHZ) will be used to target the superomedial, superolateral, and inferomedial genicular nerves, 2ml bupivacaine (0.25%) will be injected in the 3 mentioned points after a careful negative aspiration.

ELIGIBILITY:
Inclusion Criteria:

* Physical status: ASA 1 or 2 and candidates for knee arthroscopy.
* Age group: 18-50 years.
* No sex predilection.

Exclusion Criteria:

* Physical status: ASA III or above.
* Patients with a history of drug allergies to study drugs.
* Previous trauma or surgery to the leg.
* Opioids or alcohol abuse.
* Bleeding tendency.
* Dysesthesia, loss of sensation around the knee or medial aspect of the thigh.
* Inability to cooperate.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-28 (Actual); Study Completion 2024-09-28 (Actual)

PRIMARY OUTCOMES:
post-operative pain after 6 hours after the time of administration of the block according to VAS score. | During 24 hours
  * To assess postoperative pain and its intensity a segmented numeric version of the visual analogue scale (VAS) is the score that used. The patient will select a whole number (0- 10 integers) that best reflects the intensity of his pain; 1-10 is recorded by a blinded investigator during 24 hours
  * All patients receive intravenous paracetamol IV/8 hours, Patients receive intravenous pethidine 0.5mg/kg as rescue analgesia when the VAS is equal or more than 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Undecided